CLINICAL TRIAL: NCT03061773
Title: Benefits of Physical Exercise in Patients With Breast Cancer
Brief Title: Physical Training on Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Maranhao (Other)
Responsible Party: Principal Investigator, Andréa Dias Reis, Msc. Adult and Child Health and Researcher, Federal University of Maranhao
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FEDERAL UNIVERSITY OF MARANHAO
Record Dates: First submitted 2017-02-14; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Exercise group: physical training lasting 12 weeks, after detraining and in the end the control group receives physical training
  Interventions: Other: Exercise
- Group did not exercise (Active Comparator): Group did not exercise: conventional hospital treatment
  Interventions: Behavioral: Conventional hospital treatment

INTERVENTIONS:
Other: Exercise — Physical training: The combined training program consisted of 12-week aerobic, resistive and flexibility exercises, with 3 sessions per week of aerobic and resistive training in the same session (supervised by physical exercise coaches) and 2 sessions per week of Flexibility training (unsupervised). As stretching sessions were interspersed with sessions of aerobic and weathered training in the daytime period.
  Other Names: Physical exercise
  Arms: Exercise group
Behavioral: Conventional hospital treatment — Conventional hospital treatment: The patients did not perform physical training
  Arms: Group did not exercise

SUMMARY:
The treatment of breast cancer at any given time can be through surgery, as well as adjuvant treatments (radiotherapy, chemotherapy and hormone therapy) alone or together. And with this the patient tends to lose weight, he becomes depressed, resulting in an increasingly debilitating picture. Therefore, the present study aims to investigate the relationship between physical exercise and its effects on quality of life in patients with breast cancer, those who underwent surgery for at least 6 months, patients who are still with the Tumor using the adjuvant treatments submitted to physical exercises and not submitted. The sample will consist of 25 to 50 female patients aged 18 to 75 years. Patients will be submitted to the initial quality of life evaluation (SF - 36 reduced version, Anxiety and depression (HAD Scale), Fatigue (Piper Fatigue Scale), Pain (Brief Inventory of Pain), Body Composition (Bioimpedance BYODINAMICS 450 ) And oxidative stress markers (oxidized and reduced glutathione, TBARS / MDA, Myeloperoxidase and Creatinine), inflammatory markers (IL1, IL6, IL8, IL10, MCP-1 and TNF-α), hormones Estrogen, progesterone), blood test (complete blood count) 24 hour food recall (24hs food recall), and perform the maximum repetition test to find the initial workload that will be adjusted every 4 weeks with the evaluation of the load and Completing the 12 weeks of training will be reevaluated following the initial evaluation. The data collected will be treated statistically with an α=5% using the software Stata 12.0.

DETAILED DESCRIPTION:
The patients will be allocated into two groups: exercise group (intervention) and conventional treatment group (active comparison). Intervention: The combined training program consisted of 12-week aerobic, resistive and flexibility exercises, with 3 sessions per week of aerobic and resistive training in the same session (supervised by physical exercise coaches) and 2 sessions per week of Flexibility training (unsupervised). As stretching sessions were interspersed with sessions of aerobic and weathered training in the daytime period.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients;
* Sedentary;
* Currently at treatment and clinical follow-up.

Exclusion Criteria:

* Musculoskeletal injuries or disorders;
* Mental illnesses;
* Enrolled in other exercise program.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
Measure the pain, The Brief Pain Inventory (BPI). | 12 weeks
  Reduction of pain due to increased functional capacity

SECONDARY OUTCOMES:
Measure the Fatigue; The revised piper fatigue scale (PFS-R). | 12 weeks
  Reduction of fatigue due to increased functional capacity

CONTACTS AND LOCATIONS:
Overall Officials: JOÃO BS GARCIA, Doctor, Study Director — Federal University of Maranhão

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Backman M, Wengstrom Y, Johansson B, Skoldengen I, Borjesson S, Tarnbro S, Berglund A. A randomized pilot study with daily walking during adjuvant chemotherapy for patients with breast and colorectal cancer. Acta Oncol. 2014 Apr;53(4):510-20. doi: 10.3109/0284186X.2013.873820. Epub 2014 Jan 24. PMID 24460069
- [Background] Do J, Cho Y, Jeon J. Effects of a 4-week multimodal rehabilitation program on quality of life, cardiopulmonary function, and fatigue in breast cancer patients. J Breast Cancer. 2015 Mar;18(1):87-96. doi: 10.4048/jbc.2015.18.1.87. Epub 2015 Mar 27. PMID 25834616
- [Background] Nyrop KA, Callahan LF, Rini C, Altpeter M, Hackney B, Schecher A, Wilson A, Muss HB. Adaptation of an Evidence-Based Arthritis Program for Breast Cancer Survivors on Aromatase Inhibitor Therapy Who Experience Joint Pain. Prev Chronic Dis. 2015 Jun 11;12:E91. doi: 10.5888/pcd12.140535. PMID 26068412
- [Background] Sullivan AB, Scheman J, Venesy D, Davin S. The role of exercise and types of exercise in the rehabilitation of chronic pain: specific or nonspecific benefits. Curr Pain Headache Rep. 2012 Apr;16(2):153-61. doi: 10.1007/s11916-012-0245-3. PMID 22258395
- [Background] Travier N, Velthuis MJ, Steins Bisschop CN, van den Buijs B, Monninkhof EM, Backx F, Los M, Erdkamp F, Bloemendal HJ, Rodenhuis C, de Roos MA, Verhaar M, ten Bokkel Huinink D, van der Wall E, Peeters PH, May AM. Effects of an 18-week exercise programme started early during breast cancer treatment: a randomised controlled trial. BMC Med. 2015 Jun 8;13:121. doi: 10.1186/s12916-015-0362-z. PMID 26050790
- [Derived] Reis AD, Pereira PTVT, Diniz RR, de Castro Filha JGL, Dos Santos AM, Ramallo BT, Filho FAA, Navarro F, Garcia JBS. Effect of exercise on pain and functional capacity in breast cancer patients. Health Qual Life Outcomes. 2018 Apr 6;16(1):58. doi: 10.1186/s12955-018-0882-2. PMID 29625622